CLINICAL TRIAL: NCT04882189
Title: A Prospective Randomized Controlled Masked Study of Endothelial Cell Condition After Cataract Surgery Performed Using Manual Capsulorhexis or the ZEPTO Precision Capsulotomy System
Brief Title: Study of Endothelial Cell Condition After Cataract Surgery Performed Using Capsulorhexis or ZEPTO
Acronym: ZEPTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centricity Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13803
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Endothelial Cell Density Loss
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Capsulorhexis: Capsulotomies conducted by Capsulorhexis
  Interventions: Diagnostic Test: Imaging
- ZEPTO Precision Capsulotomy Device: Capsulotomies conducted by ZEPTO Precision Capsulotomy Device
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — Images of the corneal endothelium will be obtained using specular microscopy at 1- and 3-months post cataract surgery.

SUMMARY:
This study will use images of the subjects' corneal endothelium obtained using non-invasive specular microscopy to obtain corneal endothelial cell density, the coefficient of variation in endothelial cell size, and the percentage of hexagonal endothelial cells following routine cataract surgery performed using the standard method of manual capsulorhexis compared to cataract surgery performed using Zepto Precision Capsulotomy System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects consenting to undergoing phacoemulsification and IOL implant surgery for the treatment of symptomatic age-related lens cataract, and then electing to undergo the study,
* Subjects must be willing and able to return for scheduled treatment and follow-up examinations at 1 and 3 months.

Exclusion Criteria:

* Pre-existing corneal endothelium pathology
* Presence of guttae
* Narrow angle glaucoma or advanced glaucoma
* Psuedoexfoliation
* Zonular abnormalities
* Corneal endothelial cell density less than 1800 cells/mm2
* Uveitis
* Anterior chamber depth less than 2.5mm or greater than 3.75mm
* Cataract grade LOCS II > 3
* Posterior polar cataract
* Planned implantation of IOL > 25D
* Prior ocular surgery in the study eye
* History of medications with potential corneal endothelial cell toxicity
* Any condition that in the surgeon's judgement should exclude the subject from study enrollment.
* Current participation in another drug or device clinical study, or participation in such a clinical study within the prior six months and during the duration of the current study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with symptomatic age-related lens cataract desiring lens extraction and IOL implantation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Endothelial Cell Density Loss | 3 months
  Post Cataract Surgery

SECONDARY OUTCOMES:
Endothelial Cell Density Loss | 1 month
  Post Cataract Surgery
Coefficient of Variation in Endothelial Cell Size | 1 and 3 months
  Post Cataract Surgery
% of hexagonal cells | 1 and 3 months
  Post Cataract Surgery

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UltraVision, Eagle Pass, Texas
  - Houston Eye Associates, Houston, Texas
  - UltraVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided